CLINICAL TRIAL: NCT06118775
Title: Assessment of the Effectiveness and Safety of Dynamic Arterial Elastance in Weaning Vasopressor Support in Patients with Septic Shock: a Randomized Controlled Clinical Trial At Santa Fé Foundation in Bogotá
Brief Title: Evaluating Dynamic Arterial Elastance in Septic Shock Patients.
Acronym: EaDyn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Jorge Iván Alvarado, Anesthesiologist, Fundación Santa Fe de Bogota
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SECEC-2023-123
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Septic Shock
Keywords: Dynamic arterial elastance (EaDyn).; vasopressor weaning.; septic shock.
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: An open-label, pragmatic, parallel-group, controlled clinical trial will be conducted with two patient groups. Our hypothesis is that using EaDyn as a hemodynamic tool to guide vasopressor weaning can reduce the duration of vasopressor support. Patients meeting the inclusion criteria will be randomly assigned to one of the two groups using computer-generated random numbers in a 1:1 ratio. In the first group, termed 'EaDyn weaning arm' (EaDyn), dynamic arterial elastance will be used as a tool for vasopressor weaning. In the second group, named 'PAM weaning arm,' mean arterial pressure will be used as the tool for vasopressor weaning. Due to the study's methodological characteristics, blinding of participants and investigators regarding group assignment will not be possible. Lastly, the study will be conducted on an intention-to-treat basis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EaDyn weaning arm (Experimental): In the EaDyn weaning arm of the study, dynamic arterial elastance (EaDyn) will be utilized as a specialized hemodynamic tool to guide the gradual reduction of vasopressor support in patients diagnosed with septic shock. EaDyn, a measure of the relationship between arterial pressure and stroke volume variation over the cardiac cycle, provides valuable insights into vascular tone and cardiac performance
  Interventions: Procedure: EaDyn Weaning Arm:
- PAM weaning arm (Active Comparator): In the PAM (Mean Arterial Pressure) weaning arm of the study, mean arterial pressure (MAP) will be used as the primary parameter to guide the gradual reduction of vasopressor support in patients diagnosed with septic shock. Mean arterial pressure represents the average pressure in the arteries during one cardiac cycle and is a crucial indicator of perfusion to vital organs. Participants in this group will be monitored continuously for their MAP values, allowing real-time assessment of their hemodynamic status.
  Interventions: Procedure: PAM Weaning Arm:

INTERVENTIONS:
Procedure: EaDyn Weaning Arm: — The initiation of vasopressor weaning coincides with the beginning of the stabilization phase, which occurs when patients achieve a MAP >75 mmHg, a cardiac index (CI) >2.5 L/min/m², and a lactate level <2 mmol/L. The norepinephrine dose will be gradually tapered, decreasing by 0.02 mcg/kg/min every 30 minutes. In the experimental group, vasopressor weaning is guided by the EaDyn value. Weaning can proceed as long as the EaDyn remains at or above 0.90. However, if the value drops below 0.90, the weaning process halts, and the norepinephrine dose is reverted to the last dose where the EaDyn value was ≥ 0.90. Regardless of the EaDyn value, any patient experiencing a MAP decline below 50 mmHg will be withdrawn from the study. Should the MAP range between 50 mmHg and 69 mmHg, a fluid challenge of 250 mL of isotonic crystalloid must be administered before weaning continues.
  Arms: EaDyn weaning arm
Procedure: PAM Weaning Arm: — The initiation of vasopressor weaning coincides with the beginning of the stabilization phase, which occurs when patients achieve a MAP >75 mmHg, a cardiac index (CI) >2.5 L/min/m², and a lactate level <2 mmol/L. The norepinephrine dose will be gradually tapered, decreasing by 0.02 mcg/kg/min every 30 minutes. In the control group, vasopressor weaning progresses as long as the MAP remains at or above 70 mmHg. If the MAP falls between 50 and 69 mmHg, preload dependency is reassessed. Upon confirmation, a new fluid challenge is administered; vasopressor weaning halts, and the vasopressor dose reverts to its prior value. The weaning process can continue as long as the patient's MAP remains above 50 mmHg. If the MAP drops below this threshold, the patient exits the study.
  Arms: PAM weaning arm

SUMMARY:
Assess the effectiveness and safety of using dynamic arterial elastance as a tool for weaning vasopressor support in patients with septic shock, compared to a control group

DETAILED DESCRIPTION:
An open-label, randomized controlled clinical trial will be conducted with two patient groups. Our hypothesis is that using dynamic arterial elastance (EaDyn) as a tool to guide vasopressor weaning can reduce the duration of vasopressor support. Eligible patients will be randomly assigned to either the EaDyn weaning arm or the mean arterial pressure (MAP) weaning arm in a 1:1 ratio. Blinding of participants and investigators will not be possible due to the study's methodology. The analysis will be conducted on an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Admission to the ICU.
* Septic shock defined according to the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3).
* Hypotension requiring vasopressor support to maintain a MAP ≥ 65 mmHg.
* SOFA score ≥ 4.
* Vasopressor support duration ≥ 4 hours.
* Patients requiring mechanical ventilation.
* Patients who have reached the hemodynamic stabilization phase and are ready to begin the vasopressor weaning process with norepinephrine, defined as: mean arterial pressure (MAP) > 75 mmHg, cardiac index (CI) > 2.5 L/min/m², and lactate level < 2 mmol/L.

Exclusion Criteria:

* Pregnant individuals.
* Hemodynamic instability due to cardiac arrhythmias.
* Hepatic cirrhosis.
* Kidney or liver transplant.
* High probability of mortality within 24 hours, according to medical judgment.
* Left ventricular ejection fraction (LVEF) less than 50%.
* Right ventricular dysfunction, defined as a TAPSE (Tricuspid Annular Plane Systolic Excursion) measurement of less than 1.6 cm.
* Patients spontaneously breathing.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Duration of vasopressor support | 30 days
  Defined as the time interval in hours from the initiation of vasopressor support to its discontinuation.

SECONDARY OUTCOMES:
Cumulative vasopressor dosage. | 30 days
  Total dose of norepinephrine administered from the initiation of vasopressor support to its discontinuation.
Overall hospital length of stay in days | 90 days
  Length of stay in the hospital in days.
Overall ICU length of stay in days. | 90 days.
  Length of stay in the intensive care unit (ICU) in days.
Acute Kidney Injury (AKI). | 90 days.
  Proportion of AKI assessed according to the Kidney Disease Improving Global Outcomes (KDIGO) guidelines.
Mortality | 90 days.
  The number or percentage of deaths among patients diagnosed with septic shock during their hospitalization period.

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge Iván Alvarad, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarado Sanchez JI, Montanez-Narino AV, Cardenas-Bolivar YR, Stozitzky-Rios MV, Mora-Salamanca AF. Efficacy and safety of dynamic arterial elastance for weaning vasopressor support in septic shock patients: a randomised controlled trial protocol. BMJ Open. 2024 Aug 7;14(8):e086388. doi: 10.1136/bmjopen-2024-086388. PMID 39117412